CLINICAL TRIAL: NCT03665441
Title: A Randomized, Phase 3 Study of Eryaspase in Combination With Chemotherapy Versus Chemotherapy Alone as 2nd-Line Treatment of Patients With Pancreatic Adenocarcinoma
Brief Title: Study of Eryaspase in Combination With Chemotherapy Versus Chemotherapy Alone as 2nd-Line Treatment in PAC
Acronym: Trybeca-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ERYtech Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRASPANC 2018-01
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2021-01

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: pancreatic; cancer; asparaginase; gemcitabine; Abraxane; asparagine depletion; onivyde; nab-paclitaxel; folinic acid; fluorouracil; irinotecan; leucovorin; amino acid; RECIST 1.1
MeSH Terms: conditions — Neoplasms | interventions — eryaspase; Asparaginase; Gemcitabine; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Paclitaxel; Irinotecan; Fluorouracil; Leucovorin; irinotecan sucrosofate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eryaspase plus Chemotherapy (Experimental): eryaspase 100 U/kg dosed every 2 weeks in combination with
  Gemcitabine plus abraxane (albumin-bound paclitaxel) administered on Days 1, 8, and 15 of each 4 week cycle as follows:
  * Abraxane (125 mg/m2) IV
  * Gemcitabine (1000 mg/m2) IV
  Or
  Irinotecan plus 5-FU plus leucovorin administered on Days 1 and 15 of each 4 week cycle as follows:
  * Onivyde 70 mg/m2 (irinotecan freebase) IV (recommended dose in patients homozygous for UGT1A1*28 is 50 mg/m2)
  * Leucovorin 400 mg/m2 IV
  * 5 FU 2400 mg/m2
  Or
  * FOLFIRI: Irinotecan 180 mg/m2 IV
  * Leucovorin 400 mg/m² IV
  * 5 FU 400 mg/m² IV bolus
  * 5 FU 2400 mg/m² IV continuous infusion over 46 hours immediately following bolus 5 FU
  Interventions: Drug: eryaspase; Drug: Gemcitabine plus Abraxane; Drug: Irinotecan plus 5-FU plus leucovorin
- Chemotherapy alone (Other): Standard treatment: Gemcitabine plus abraxane (albumin-bound paclitaxel) administered on Days 1, 8, and 15 of each 4 week cycle Or Irinotecan plus 5-FU plus leucovorin administered on Days 1 and 15 of each 4 week cycle
  Interventions: Drug: Gemcitabine plus Abraxane; Drug: Irinotecan plus 5-FU plus leucovorin

INTERVENTIONS:
Drug: eryaspase — L-asparaginase encapsulated in erythrocytes (red blood cells)
  Other Names: L-asparaginase
  Arms: Eryaspase plus Chemotherapy
Drug: Gemcitabine plus Abraxane — gemcitabine, Abraxane
  Other Names: Gemzar, nab-paclitaxel, onxol
Drug: Irinotecan plus 5-FU plus leucovorin — irinotecan, 5-FU, leucovorin
  Other Names: Onivyde, liposomal irinotecan, Camptosar, Campto, Adrucil, Carac, Efudex, Efudix, folinic acid, calcium folinate

SUMMARY:
This is an open-label, multicenter, randomized, Phase 3 study in patients with ductal adenocarcinoma of the pancreas who have failed only one prior line of systemic anti-cancer therapy for advanced pancreatic cancer and have measurable disease.

DETAILED DESCRIPTION:
Patients who meet all inclusion and exclusion criteria will be randomized in a 1:1 ratio to one of the following treatment arms (see figure below):

* Arm A (investigational arm): eryaspase in combination with either gemcitabine/Abraxane or irinotecan-based therapy (FOLFIRI [FOLinic acid-Fluorouracil-IRInotecan regimen] or Onivyde®/5 fluorouracil/leucovorin), or
* Arm B (control arm): gemcitabine/Abraxane or irinotecan-based therapy (FOLFIRI or Onivyde/5-FU/leucovorin)

The chemotherapy will be investigator's choice and based on what patient has received in first line treatment. Treatment will continue until disease progression, unacceptable toxicity, or the patient's withdrawal of consent.

An End of Treatment visit should occur within approximately 30 days from last dose of eryaspase or chemotherapy regimen.

A survival follow-up period will include the collection of survival, progression of disease if applicable, treatment updates, and quality of life assessments every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for the study if all the following criteria are met:

1. Must be 18 years of age or older.
2. Must have histologically confirmed pancreatic adenocarcinoma.
3. Must have Stage III or IV disease.
4. Must have received one line of systemic chemotherapy in the advanced setting with or without targeted agents, immunotherapy, or radiotherapy for treatment of advanced pancreatic adenocarcinoma.
5. Must have radiological evidence of disease progression following most recent prior treatment, defined as appearance of any new lesion or increase of >20% of one or more existing lesions.
6. Must have measurable lesion(s) per RECIST version 1.1 by CT scan with contrast (or MRI, if the patient is allergic to CT contrast media).

   NOTE: Bone disease consisting of blastic lesion only is not measurable.
7. Archival or fresh tumor tissue must be available for evaluating relevant biomarkers. Formalin-fixed paraffin-embedded [FFPE] block preferred, or a minimum of 10 unstained FFPE slides of one archived block is required.

   NOTE: Cytology samples from fine needle aspirates or brushing biopsies are not sufficient.

   If archival tissue is unavailable and an elective biopsy can't be scheduled due to COVID, this will be waived.
8. Must have adequate performance status:

   1. ECOG Performance Status (PS) score of 0, or
   2. ECOG PS score one and score ≥80 on Karnofsky Performance Status (KPS) scale. NOTE: Must have body mass index (BMI) ≥18.5 kg/m2 (obtained <14 days prior to randomization.
9. Must have life expectancy of >12 weeks according to the investigator's clinical judgment.
10. Females of childbearing potential must have a negative pregnancy test at screening and additional negative pregnancy test prior to first dose. Males and females of childbearing potential must agree to use a highly effective method of contraception during treatment and for at least 6 months after the last dose of study treatment.
11. Must have adequate laboratory parameters at baseline (obtained <14 days prior to randomization). Laboratory parameters outside of these ranges that are deemed clinically insignificant should be discussed with the medical monitor:

    1. Absolute neutrophil count ≥1.5 x 109/L.
    2. Hemoglobin ≥9 g/dL. Patients with a baseline Hemoglobin ≥13 g/dL should be discussed with the medical monitor.
    3. Platelet count ≥100,000/mm3 (100 x 109/L).
    4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN) (≤5 x ULN in presence of liver metastases).
    5. Total bilirubin ≤ 1.5 x institutional ULN.
    6. Serum creatinine within normal limits or calculated clearance >60 mL/min/1.73 m2 for patients with serum creatinine levels above or below the institutional normal range.
    7. Acceptable coagulation parameters: plasma antithrombin III >70% and fibrinogen ≥1.5 g/L
    8. Serum albumin ≥3.0 g/dL.
12. Patients requiring biliary stent placement must have the biliary stent placed >7 days prior to screening and must have normalization of bilirubin level after stenting.
13. Must not be receiving therapy in a concurrent clinical study and must agree not to participate in any other interventional clinical studies during their participation in this trial while on study treatment. Patients taking part in surveys or observational studies are eligible to participate in this study.
14. Must be able to understand and comply with the conditions of the protocol and must have read and understood the consent form and provided written informed consent.

Exclusion Criteria:

A patient is not eligible to participate in the study if any of the following criteria are met:

1. Resectable or borderline resectable pancreatic adenocarcinoma at the time of signing the informed consent.
2. Histology other than pancreatic adenocarcinoma (for example, but not inclusive: neuroendocrine, adenosquamous, etc.).
3. More than one line of prior treatment in advanced or metastatic setting.
4. Patient has experienced medically significant acute decline in clinical status including

   1. Decline in ECOG PS to >1 (or KPS <70) between baseline visit and within 72 hours prior to randomization.
   2. Weight loss of ≥10% during screening.
5. Presence of active or symptomatic untreated central nervous system (CNS) metastases.

   NOTE: Patients with asymptomatic or stable CNS metastases are eligible, provided that the CNS metastases are radiologically and clinically stable, and the patient is off high-dose steroid treatment for at least one month prior to randomization.
6. Prior radiotherapy to the only area of measurable disease. NOTE: Patients must have completed treatment and recovered from all acute treatment-related toxicities prior to administration of the first dose of eryaspase or chemotherapy.
7. Bone as the only site of metastatic disease from pancreatic cancer (bone only disease).
8. History of recent clinical pancreatitis, according to revised Atlanta criteria, within 3 months of randomization.

   NOTE: The revised Atlanta classification [1] requires that two or more of the following criteria be met for the diagnosis of acute pancreatitis: (a) abdominal pain suggestive of pancreatitis, (b) serum amylase or lipase level ≥3 x ULN, or (c) characteristic imaging findings using CT or MRI.
9. Neurosensory neuropathy > Grade 2 at baseline.
10. Pregnancy or breastfeeding.
11. History of infection with human immunodeficiency virus (HIV) and/or active infection with hepatitis B or hepatitis C.

    NOTE: Patients with unknown status of hepatitis B or C must be tested and declared negative before randomization.
12. Hypersensitivity to any of the components of the chemotherapy or ASNase.
13. Patients who have received live or live attenuated vaccines within 3 weeks of randomization.
14. History of other malignancies NOTE: Adequately treated non-melanoma skin cancer or curatively treated in-situ cancer of the cervix may be eligible.

    NOTE: Patients successfully treated for other malignancies and are disease-free for at least 5 years may be eligible.
15. Any other severe acute or chronic condition/treatments that may increase the risk of study participation including:

    1. History of abdominal fistula, gastrointestinal perforation, peptic ulcer, or intra-abdominal abscess within 6 months prior to randomization.
    2. Current or history within 6 months prior to randomization of medically significant cardiovascular disease including symptomatic congestive heart failure >New York Heart Association (NYHA) Class II, unstable angina pectoris, clinically significant cardiac arrhythmia.
    3. Patients with pre-existing coagulopathy (e.g. hemophilia).
    4. Psychiatric illness/social situations or any other serious uncontrolled medical disorders in the opinion of the Investigator that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, MD, PhD, Principal Investigator — Weill Cornell, NY, US; Pascal Hammel, MD, PhD, Principal Investigator — Hospital Beaujon, Clichy, France
Locations (16):
- United States (14):
  - Arizona Cancer Center, Scottsdale, Arizona
  - St. Joseph Heritage Healthcare, Fullerton, California
  - University of California Davis Medical Center, Sacramento, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota Health Clinics and Surgery Center, Minneapolis, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University, Stony Brook, New York
  - Duke University, Durham, North Carolina
  - Medical Oncology Associates, Spokane, Washington
- Institut de Cancerologie, Brest, France
- Hammersmith Hospital, London, United Kingdom

REFERENCES:
- [Derived] Hammel P, Metges JP, Macarulla Mercade T, Garcia-Carbonero R, Bouche O, Portales F, Pazo Cid RA, Mineur L, Cubillo Gracian A, Trouilloud I, Guimbaud R, Tougeron D, Reina JJ, Feliu J, Sauri T, Fountzilas C, Lecomte T, Molin Y, Ponz-Sarvise M, Forget F, Berardi R, Van Cutsem E, Gelsomino F, Tournigand C, Bockorny B, Bachet JB, Marin Vera M, Cuyle PJ, Wasan H, Noel M, Van Laethem JL, Kay R, Youssoufian H, El-Hariry I, Hidalgo M. TRYBECA-1: A Randomized Phase III Study of Eryaspase Combined With Chemotherapy Versus Chemotherapy as Second-Line Treatment in Patients With Advanced Pancreatic Adenocarcinoma. J Clin Oncol. 2025 Dec 10;43(35):3714-3727. doi: 10.1200/JCO-25-00872. Epub 2025 Nov 4. PMID 41187298

RESULTS

PARTICIPANT FLOW:
Groups:
- Eryaspase Plus Chemotherapy: eryaspase 100 U/kg dosed every 2 weeks in combination with
  Gemcitabine plus abraxane (albumin-bound paclitaxel) administered on Days 1, 8, and 15 of each 4 week cycle as follows:
  * Abraxane (125 mg/m2) IV
  * Gemcitabine (1000 mg/m2) IV
  Or
  Irinotecan plus 5-FU plus leucovorin administered on Days 1 and 15 of each 4 week cycle as follows:
  * Onivyde 70 mg/m2 (irinotecan freebase) IV (recommended dose in patients homozygous for UGT1A1*28 is 50 mg/m2)
  * Leucovorin 400 mg/m2 IV
  * 5 FU 2400 mg/m2
  Or
  * FOLFIRI: Irinotecan 180 mg/m2 IV
  * Leucovorin 400 mg/m² IV
  * 5 FU 400 mg/m² IV bolus
  * 5 FU 2400 mg/m² IV continuous infusion over 46 hours immediately following bolus 5 FU
  eryaspase: L-asparaginase encapsulated in erythrocytes (red blood cells)
  Gemcitabine plus Abraxane: gemcitabine, Abraxane
  Irinotecan plus 5-FU plus leucovorin: irinotecan, 5-FU, leucovorin
Period: Overall Study
Arm/Group | Eryaspase Plus Chemotherapy | Chemotherapy Alone
Started | 255 | 257
Completed | 216 | 240
Not Completed | 39 | 17
Not completed — survival follow up ongoing | 23 | 0
Not completed — Patients ongoing on treatment | 9 | 6
Not completed — Randomized but not treated | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eryaspase Plus Chemotherapy | Chemotherapy Alone | Total
Number analyzed (Participants) | 255 | 257 | 512
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 140 | 142 | 282
  >=65 years | 115 | 115 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (10.29) | 62.5 (9.72) | 62.2 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 124 | 245
  Male | 134 | 133 | 267
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 235 | 248 | 483
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 5 | 17
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39
  Europe | 236 | 237 | 473
ECOG PS [Number; unit: participants] — ECOG Performance Status (PS) assesses patient's level of functioning Grade 0 to 4 in terms of their ability to care for themselves, daily activity, and physical ability:
  Grade 0=Fully active, able to carry on all pre-disease performance without restriction; Grade 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Patients with Grades 2 to 5 were not included.
  participants
    ECOG 0 | 107 | 105 | 212
    ECOG 1 | 148 | 152 | 300
Time from initial diagnosis of advanced disease to randomization [Count of Participants; unit: Participants]
  <6 months | 79 | 74 | 153
  >=6 months | 176 | 183 | 359

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: To determine whether the addition of eryaspase to chemotherapy improves OS when compared to chemotherapy alone
Time Frame: ~12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Eryaspase Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 255 | 257
months | 7.5 [6.5 to 8.3] | 6.7 [5.4 to 7.5]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: To compare PFS between the 2 treatment arm. Progression is determined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: ~24 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Eryaspase Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 255 | 257
months | 3.7 [3.4 to 4.1] | 3.4 [2 to 3.7]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: To compare the ORR between the 2 treatment arms. ORR is defined as the proportion of patients who achieve objective tumor response (CR or PR) per modified RECIST 1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: ~24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Eryaspase Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 255 | 257
Participants | 41 | 32

4. Secondary Outcome: Duration of Response (DoR)
Description: To compare the DoR between the 2 treatment arms
Time Frame: ~24 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Eryaspase Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 255 | 257
months | 5.7 [3.9 to 7.4] | 6.8 [2.8 to 7.4]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: To compare the between the 2 treatment arms
Time Frame: ~24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Eryaspase Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 255 | 257
Participants | 147 | 126

6. Secondary Outcome: Incidence of Treatment Emergent Adverse Events as Assessed by CTCAE v5.0
Description: To evaluate the safety and tolerability of eryaspase in combination with chemotherapy versus chemotherapy alone by assessing the number of patients with with treatment emergent adverse events per CTCAE v5.0
Time Frame: ~9 months
Population: Analysis set includes only patients who were treated on study (Safety Population). 7 patients in the eryaspase plus chemotherapy arm and 11 patients in the chemotherapy alone arm discontinued study prior to initiation of first dose.
Measure: Number; unit: participants
Arm/Group | Eryaspase Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 248 | 246
participants
  Number of patients with treatment emergent adverse events (TEAE) | 248 | 246
  number of patients with TEAE >= Grade 3 | 195 | 176
  Number of patients with TE SAE | 122 | 105
  Number of patients with TEAEs leading to study drug discontinuation | 46 | 41
  Number of patients with TE SAE with outcome of death | 14 | 9

7. Secondary Outcome: Time to Quality of Life Questionnaire EORTC QLQ-C30 First Worsening in Global Health Status Analysis
Description: The time to first Worsening was defined as the date of randomization to the date of first Worsening occurred in patient score on their global health status. Patients who did not have any worsening were censored at date of last measurement or at baseline if no measurement is available post-baseline.
Time Frame: ~1 year
Population: The number of participants in this section consist of all patients who receive at least one dose of the study treatment and provide answers to at least some items of the EORTC QLQ-C30 at Cycle 1 Day 1 (i.e, baseline) and a time point after the date of first dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Eryaspase Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 228 | 229
months | 4.0 [3.1 to 5.1] | 3.6 [2.8 to 4.7]

ADVERSE EVENTS:
Time Frame: 9 months (Adverse events were monitored for approximately 9 months and mortality assessed for approximately 12 months.)
Arm/Group | Eryaspase Plus Chemotherapy | Chemotherapy Alone
All-Cause Mortality (participants affected / at risk) | 209/248 | 211/246
Serious Adverse Events (participants affected / at risk) | 122/248 | 105/246
Other Adverse Events (participants affected / at risk) | 248/248 | 244/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eryaspase Plus Chemotherapy (N=248) | Chemotherapy Alone (N=246)
Gastrointestinal obstruction (Gastrointestinal disorders) | 9 | 11
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 9
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Abdominal pain (Gastrointestinal disorders) | 6 | 4
vomiting (Gastrointestinal disorders) | 3 | 2
Colitis (Gastrointestinal disorders) | 2 | 2
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Oral disorder (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1
Gastric varices (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatic duct stenosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 11 | 6
Device related infection (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 4 | 0
Bacteraemia (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Aeromonas infection (Infections and infestations) | 2 | 0
Atypical pneumonia (Infections and infestations) | 2 | 0
COVID-19 (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 1 | 1
Liver abscess (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 2
Abdominal abscess (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Interverterbral discitis (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Perihepatic abscess (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Superinfection (Infections and infestations) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 13 | 5
Bile duct stenosis (Hepatobiliary disorders) | 2 | 1
Cholestasis (Hepatobiliary disorders) | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 2
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Pyrexia (General disorders) | 10 | 6
General physical health (General disorders) | 7 | 4
Asthenia (General disorders) | 1 | 1
Inadequate analgesia (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3
Pancytopenia (Blood and lymphatic system disorders) | 4 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 | 1
Hemolytic uraemic syndrome (Blood and lymphatic system disorders) | 2 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Myelosuppression (Blood and lymphatic system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 5
Ischaemic stroke (Nervous system disorders) | 4 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Haemolytic transfusion (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Device malfunction (Product Issues) | 3 | 4
Cardiac failure (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Alloimmunisation (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Pancreatic enzymes abnormal (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eryaspase Plus Chemotherapy (N=248) | Chemotherapy Alone (N=246)
Asthenia (General disorders) | 186 | 73
Diarrhoea (Gastrointestinal disorders) | 132 | 107
Anaemia (Blood and lymphatic system disorders) | 128 | 97
Nausea (Gastrointestinal disorders) | 132 | 89
Neutropenia (Blood and lymphatic system disorders) | 108 | 93
Abdominal pain (Gastrointestinal disorders) | 96 | 84
Thrombocytopenia (Blood and lymphatic system disorders) | 75 | 72
Pyrexia (General disorders) | 73 | 56
Decreased appetite (Gastrointestinal disorders) | 77 | 62
Neuropathy peripheral (Nervous system disorders) | 69 | 62
Constipation (Gastrointestinal disorders) | 69 | 62
Vomiting (Gastrointestinal disorders) | 69 | 57
Oral disorder (Gastrointestinal disorders) | 58 | 60
Alopecia (Skin and subcutaneous tissue disorders) | 64 | 51
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 24
Hypokalaemia (Metabolism and nutrition disorders) | 29 | 26
Weight decreased (Investigations) | 35 | 14
Oedema (General disorders) | 65 | 47
Transaminases increased (Investigations) | 30 | 18
Leukopenia (Blood and lymphatic system disorders) | 28 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 21
Headache (Nervous system disorders) | 29 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 25 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 | 16
Sleep disorder (Psychiatric disorders) | 16 | 19
Dysgeusia (Nervous system disorders) | 20 | 14
Blood albumin decreased (Investigations) | 15 | 16
Hyperbilirubinaemia (Hepatobiliary disorders) | 18 | 10
Gamma-glutamyltransferase increased (Investigations) | 16 | 13
Lymphopenia (Blood and lymphatic system disorders) | 19 | 10
Rash (Skin and subcutaneous tissue disorders) | 18 | 10
Urinary tract infection (Infections and infestations) | 13 | 15
Flatulence (Gastrointestinal disorders) | 19 | 8
Anxiety (Psychiatric disorders) | 13 | 13
Blood alkaline phosphatase increased (Investigations) | 15 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 11
General physical health deterioration (General disorders) | 17 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 13
Chills (General disorders) | 17 | 6
Ascites (Gastrointestinal disorders) | 15 | 7
Dizziness (Nervous system disorders) | 12 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 10
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 12 | 10
Gastroesophageal reflux (Gastrointestinal disorders) | 15 | 6
Dyspepsia (Gastrointestinal disorders) | 12 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has rights to the first publication for up to 18 months after study completion or termination, or until sponsor determines it does not plan to publish the study results.

Following this the Institution and/or Principal Investigator may publish data or results generated at Institution; provided, the proposed publication or presentation is submitted to the Sponsor at least 45 days prior to the date of the proposed publication or presentation for review and approval.

DOCUMENTS (2):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03665441/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03665441/SAP_001.pdf